CLINICAL TRIAL: NCT00898599
Title: Investigation of the Effects of a Prebiotic Supplement on Immune Function in Healthy Human Adults
Brief Title: Prebiotics and Immune Function in Middle Aged Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RHMNUT0055
Record Dates: First submitted 2009-04-20; First posted 2009-05-12 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2010-07

CONDITIONS: Immune Function
MeSH Terms: interventions — Prebiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Prebiotic (Experimental): Inulin type fructooligosaccharides
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Inulin type fructooligosaccharides
  Other Names: Synergy1
  Arms: Prebiotic
Dietary Supplement: Placebo — Maltodextrin as placebo
  Other Names: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
Prebiotics are naturally occurring carbohydrates found in a variety of edible plants. They are not digested by mammalian enzymes, and so reach the gut intact, where they are fermented by some species of intestinal bacteria. This fermentation is thought to have several benefits for the host including improving immune function. There are numerous methods available for assessing the human immune response. Response to vaccination is thought to be a good method for this. Not many studies have examined the effect of prebiotics on the human immune response to vaccination. Thus the investigators propose to test the effect of a prebiotic on the immune response in healthy volunteers including their response to the current flu vaccine. The investigators hypothesise that the prebiotic will enhance the immune response including the response to the vaccine.

DETAILED DESCRIPTION:
Prebiotics are naturally occurring carbohydrates found in a variety of edible plants. They are not digested by mammalian enzymes, and so reach the gut intact, where they are fermented by some species of intestinal bacteria. This fermentation is thought to have several benefits for the host including improving the immune response. Inulin-type fructans (oligofructose and inulin) are classified as prebiotics. Inulin is found naturally in significant amounts in a variety of plants foods, such as bananas, leeks, onions, artichokes, wheat and chicory. Synergy1 is a prebiotic preparation produced by Beneo-Orafti, and containing a mixture of oligofructose and inulin derived from chicory. Fructooligosaccharides including Synergy1 are widely used by the food industry and are commonly found as a source of insoluble fibre in many biscuit, bakery, cereal and dairy products.

There is increasing evidence that the changes in the intestinal microflora that occur with the consumption of fructooligosaccharides can modulate immune parameters, not only in the gut-associated lymphoid tissue, but also secondary lymphoid tissues and the peripheral circulation. Much of the evidence for beneficial effects of fructooligosaccharides on immune function comes from animal models e.g. rats, mice, dogs and pigs. Results from these studies show that the innate and adaptive immune systems of both the gut associated lymphoid tissue and the systemic immune system can be modified by fructooligosaccharides. However, there are few human studies so far which have investigated the effects of prebiotics on immune function, and these studies mostly rely on systemic markers of immunity. The results show little effect of fructooligosaccharides on innate immune function, but mixed results are reported regarding the adaptive immune system, suggesting that there may by improvement on this aspect of immunity with increased intake of fructooligosaccharides. The small number of published human studies led Watzl et al. (2005) to suggest that more human studies are needed to find out whether inulin and/or oligofructose have the potential to modulate systemic immunity in well-nourished individuals.

There are numerous methods available for assessing the human immune response. These have been evaluated by a panel of European experts (Albers et al. 2005). Based on its biological relevance, sensitivity and practical feasibility, response to vaccination was identified by this panel as the gold standard for measuring the functioning of the immune system in vivo (Albers et al. 2005). A small number of studies have studied the effect of fructooligosaccharides on the human immune response using vaccination response as the outcome, but only four of these examined fructooligosaccharides in the absence of other additional nutrients and of these two studies were in infants. Thus, the number of studies examining the immunologic impact of fructooligosaccharides in adult humans and using the gold standard outcome is very limited. From a public health perspective, it would be of importance, if fructooligosaccharides can improve immune function especially in older adults who are at risk of age-related immune decline. Thus, we propose to use a commercially available influenza vaccine (Imuvac®) to stimulate the immune response in healthy human adults, and to use this to assess the effect of a well defined prebiotic preparation commonly used in the food industry (Synergy1).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 45-65 years
2. Body mass index 20 to 32 kg/m2.
3. Not consuming probiotic supplements, yoghurts, drinks or other foods
4. Not consuming prebiotic supplemented drinks or foods
5. In general good health
6. No antibiotic use in the 2 months prior to entering the study or during the study
7. Not been vaccinated with the current season's influenza vaccine
8. Being able to provide written informed consent

Exclusion Criteria:

1. Aged < 45 or > 66 years
2. Body mass index < 20 or > 32 kg/m2.
3. Being diabetic (type 1 or type 2)
4. Displaying manifestations of allergy - asthma, hay-fever, dermatitis - or being treated for these
5. Being egg allergic
6. Use of any prescribed medicine (unless deemed to be acceptable by the PI)
7. Suffering from any infectious illness
8. Chronic gastrointestinal problems (e.g. IBD, IBS, cancer)
9. Recent blood donation
10. Participation in another clinical trial
11. Use of prebiotic or probiotic supplements, foods or drinks
12. Consuming vitamin, mineral or oil supplements
13. Previously vaccinated with the influenza vaccine being used.

Ages: 45 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Serum anti-vaccine antibody concentrations | Weeks 2 and 4 post-vaccination

SECONDARY OUTCOMES:
Serum total antibody (IgG, IgA, IgM) concentrations | Weeks -4, 0, 2 and 4 with respect to vaccination
Innate immune responses - neutrophil and monocyte phagocytosis and respiratory burst | Weeks -4, 0, 2 and 4 with respect to vaccination
Ex vivo T lymphocyte responses to mitogen (activation, proliferation and cytokine production) | Weeks -4, 0, 2 and 4 with respect to vaccination
Ex vivo T lymphocyte responses to vaccine (activation, proliferation and cytokine production) | Weeks 0, 2 and 4 with respect to vaccination
Ex vivo natural killer cell activity | Weeks -4, 0, 2 and 4 with respect to vaccination
Faecal microflora | Weeks -4 and 0 with respect to vaccination
Salivary IgA concentration | Weeks -4, 0, 2 and 4 with respect to vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Calder, PhD, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, United Kingdom